CLINICAL TRIAL: NCT03817710
Title: Prevalence of Tics in Childern With Acute Deficit Hyper Activity Syndrom
Brief Title: Tics in Childern With Acute Deficit Hyper Activity Syndrom
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Hassobba, principle investigator, Assiut University
Other Study IDs: POTIADHD
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Behavior Disorders
Keywords: tics disorder in childern with acute deficit hyper activity syndrom
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tics have been defined as sudden, rapid, recurrent, non-rhythmic, stereotyped, involuntary movements or vocalizations. Motor tic can be either simple or complex, depending on whether one or several muscle groups are simultaneously or concurrently affected. Motor tics commonly include behaviours such as eye blinking, lip-licking, or mouth opening. It can also involve more complex movements like facial grimacing ,head movements , shoulder shrugging or combinations of these.Vocal or phonic tics are involuntary sounds that include throat clearing, coughing, barking, sniffing, unnecessary belching or more complex vocalizations such as repeating parts of words or phrases.

Gilles de la Tourette's syndrome is complex neurodevelopmental disorder characterized by combination of motor and vocal tics. Motor tics often precede the onset of phonic tics by many years. The phonic tics may commence from about the age of 3 years. Severe Tourette's Syndrome may manifest as forceful bouts of self-harming motor tics, including hitting or biting, as well as socially unacceptable utterances (coprolalia) and gestures [3].

The Tourette's Syndrome Study Group definition from 1993 requires the concurrent presence of motor and vocal tics occurring almost daily for at least one year, [4]. The Diagnostic and Statistical Manual of Mental Disorders 5th Edition requires both multiple motor and one or more vocal tics have been present at some time during the illness, although not necessarily concurrently for the diagnosis of Tourette's Syndrome . It also describes Tics Disorder and Tourette's Syndrome as waxing and waning in frequency and symptoms must have lasted for more than one year since the first onset.

DETAILED DESCRIPTION:
The average age of developing Tourette's Syndrome is 7 years, with a range from three to eight years. Most patients with childhood tics disorder show remarkable symptoms improvement by the age of 19 years. Adult-onset cases of Tourette's Syndrome are usually the most severe forms of presentation...

Motor or phonic tics often begin with the patient experiencing some psycho-sensory phenomena known as the "premonitory urge" which may be localized to an area of the tics or a generalised inner tension. Most individuals with Tics/ Tourette's Syndrome also experience feelings of momentary relief after the tic has occurred. TICS Disorder are typically exacerbated by stressful life-events associated with high levels of emotional excitements and fatigue, and can include normally routine activities such as the start of school, birthdays, arrival of a new sibling, changes in the social or physical environment like moving house or going on holidays. The symptoms of childhood Tics Disorder / Tourette's Syndrome are usually mild and they are almost invariably co-morbid with other mental health and behavioural problems including ADHD, Obsessive-compulsive disorder (OCD), learning disabilities (LD) and mood disorders. Tics/ Tourette's Syndrome can significantly impair the patient's self-esteem, peer and or family relationships[3]. Although tics often improve after adolescence, recent studies suggest that comorbid OCD and ADHD often persist.

Other common comorbidities in children with Tics/ Tourette's Syndrome include anxiety disorders, depression, autistic spectrum disorder (ASD), conduct disorder (CD), oppositional defiant disorder (ODD), self-injurious behaviours, sleep disorders, rage attacks and personality disorder.

ADHD :

Attention deficit hyperactivity disorder (ADHD) is the commonest neurobehavioural disorder in children and adolescents, with prevalence ranging between 5% and 12% in the developed countries[2]. Up to 80% of ADHD patients have one or more co-morbid conditions which include Tics disorders (TD). There is a complex interplay between Tics Disorder and ADHD in children and young people. TDs are common comorbidities in paediatric ADHD patients with or without treatment with pharmacotherapy. ADHD and other co-morbid disorders like Tics/ Tourette's syndrome (TS), especially if left untreated, can have lasting impairing effects on several aspects of daily functioning. Tics naturally wax and wane in clinical severity and are exacerbated by stress, including consequences of untreated ADHD. There has been conflicting evidence of the role of psychostimulants in either precipitating or exacerbating TDs in ADHD patients. Some evidence also suggests that tics may improve with ADHD treatment Tics naturally wax and wane in clinical severity and are exacerbated by stress, including consequences of untreated ADHD. There has been conflicting evidence of the role of psychostimulants in either precipitating or exacerbating TDs in ADHD patients. Some evidence also suggests that tics may improve with ADHD treatment

ELIGIBILITY:
Inclusion Criteria:

* infants with ADHD aged between 2 and 18 years (old and new).

Exclusion Criteria:

* Infants below 2 or above 18 .

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All cases will subjected for full clinical history including different manifestation of tics Data were collected from (Children Hospital ) Assiut University outpatient clinics with the purpose to study tics in children with ADHD.( ADHD Score)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Tics Disorder in Children With ADHD | one year
  Prevalence of Tics Disorder in Children With ADHD

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biederman J, Faraone SV. Attention-deficit hyperactivity disorder. Lancet. 2005 Jul 16-22;366(9481):237-48. doi: 10.1016/S0140-6736(05)66915-2. PMID 16023516
- [Background] Faraone SV, Sergeant J, Gillberg C, Biederman J. The worldwide prevalence of ADHD: is it an American condition? World Psychiatry. 2003 Jun;2(2):104-13. PMID 16946911
- [Result] Anckarsater H, Lundstrom S, Kollberg L, Kerekes N, Palm C, Carlstrom E, Langstrom N, Magnusson PK, Halldner L, Bolte S, Gillberg C, Gumpert C, Rastam M, Lichtenstein P. The Child and Adolescent Twin Study in Sweden (CATSS). Twin Res Hum Genet. 2011 Dec;14(6):495-508. doi: 10.1375/twin.14.6.495. PMID 22506305
- [Result] Beau-Lejdstrom R, Douglas I, Evans SJ, Smeeth L. Latest trends in ADHD drug prescribing patterns in children in the UK: prevalence, incidence and persistence. BMJ Open. 2016 Jun 13;6(6):e010508. doi: 10.1136/bmjopen-2015-010508. PMID 27297009